CLINICAL TRIAL: NCT05837026
Title: Randomized Controlled Trial of Health System/Community Partnership for Enhanced Outreach to Prevent Suicide Attempts
Brief Title: A Health System/Community Partnership for Enhanced Outreach to Prevent Suicide Attempts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Samaritans of Boston (Unknown)
Responsible Party: Principal Investigator, Jordan W. Smoller, MD, Associate Chief for Research, Department of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023P000611-B
Record Dates: First submitted 2023-04-11; First posted 2023-05-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation
Keywords: Suicide; Suicidal Thoughts
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Effectiveness-implementation Hybrid Type 1 randomized trial. Participants will be randomized to EOI plus care as usual (CAU) or CAU alone using an equal (1:1) allocation ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Outreach Intervention plus Care as Usual (CAU) (Experimental): Participants will receive the Enhanced Outreach Intervention (EOI) plus care as usual for 12 weeks after ED discharge.
  Interventions: Behavioral: Enhanced Outreach Intervention (EOI) plus Care as Usual (CAU)
- Care as Usual (CAU) (Other): Participants will receive the standard care (i.e., CAU) that the hospital provides to patients who present with suicidal thoughts.
  Interventions: Other: Care as Usual (CAU)

INTERVENTIONS:
Behavioral: Enhanced Outreach Intervention (EOI) plus Care as Usual (CAU) — The EOI will contain four main components: safety planning, caring contacts, care engagement, and risk assessment.
  Outreach (via phone or text messaging) from Samaritans staff will be conducted every week of the 12 week intervention. Conversations will use a standardized phone script to (a) conduct a risk assessment, (b) develop and review a list of coping skills to use if the participant has suicidal thoughts, and (c) discuss plans for receiving mental health care. Samaritans staff will also send a caring text message or email at least once per week.
  Participants will also receive standard care that hospitals provide to patients who present with suicidal thoughts.
  Arms: Enhanced Outreach Intervention plus Care as Usual (CAU)
Other: Care as Usual (CAU) — Participants will receive standard care that hospitals provide to patients who present with suicidal thoughts.
  Arms: Care as Usual (CAU)

SUMMARY:
The goal of this study is to test an enhanced outreach intervention (EOI) delivered by Samaritans of Boston (a community organization that provides support during mental health crises) for people after they leave an emergency department (ED) visit for suicidal thoughts. The main questions it aims to answer are:

* Does the EOI reduce suicide-related behaviors?
* Does the EOI increase outpatient treatment attendance?
* Is the EOI acceptable and feasible?
* Can the EOI be delivered with fidelity by Samaritans?

Participants will be randomized to the EOI plus care as usual or care as usual alone. Participants in the EOI plus care as usual group will:

* Receive outreach (by call or text) at a planned time once per week for the next 12 weeks. During these conversations, Samaritans staff will ask participants questions about their suicidal thoughts and behaviors, develop and review a list of coping skills to use if they have suicidal thoughts, and discuss plans for receiving mental health care.
* Receive caring messages from Samaritans staff at least once per week.
* Receive standard care that hospitals give for patients who present with suicidal thoughts.
* Be asked to complete monthly self-report questionnaires.

For care as usual alone, participants will:

* Receive standard care that hospitals give for patients who present with suicidal thoughts.
* Be asked to complete monthly self-report questionnaires.

DETAILED DESCRIPTION:
The period after discharge from an emergency department (ED) is a critical time of increased risk for suicide and related behavior (SRB). Brief "caring contact" interventions that provide follow-up and support after a healthcare visit have been shown to reduce SRB and are now recommended best practices for suicide prevention in healthcare systems. However, system- and individual-level barriers to widespread implementation exist. For example, deployment of brief contact interventions requires dedicated resources and staffing within already overburdened healthcare settings, and even single-session interventions require robust provider training and ongoing oversight for successful implementation.

The purpose of this study is to evaluate a recently developed Enhanced Outreach Intervention (EOI) for post-ED discharge that combines multiple evidence-based suicide prevention components (e.g., safety planning, risk assessment, caring contacts, and care engagement) and is delivered through a partnership between a healthcare system (Mass General Brigham [MGB]) and a local crisis line organization (Samaritans of Boston). Combining multiple evidence-based interventions has the potential to increase effectiveness over usual practices, and partnering with a community organization vastly increases scalability.

Samaritans staff will undergo robust, multifaceted training on the EOI, and use standardized decision trees to guide EOI delivery. The investigators will conduct a randomized controlled trial (N=300) of the EOI plus care as usual versus care as usual alone after ED discharge to test effectiveness of the EOI and collect data on implementation-related factors. The investigators will also explore potential moderators of intervention effects, including age, sex, race/ethnicity, and predicted risk of suicide attempt at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Currently a patient being treated and evaluated by psychiatry service in an MGB ED
2. Participants enrolled in another study (NCT05671133; PI Nock) conducted by the research team who fall into the top 50% of risk based on the suicide risk prediction algorithm used in that study
3. Able to read English
4. Ownership of a smartphone (iOS or Android) and consistent access to their smartphone following discharge from the current treatment unit or program; ability to be reliably contacted
5. Willing to provide contact information for collateral contact
6. Willing to share contact information and key clinical information with Samaritans of Boston
7. Consent to unencrypted text or email communications
8. Willing to provide social security number (SSN) or individual taxpayer identification number (ITIN) for study compensation

Exclusion Criteria:

1. Any factor that impairs an individual's ability to comprehend and effectively participate in informed consent, including the presence of gross cognitive impairment due to florid psychosis, intellectual disability, dementia, or acute intoxication
2. Presence of extremely agitated or violent behavior at the time of consent or enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of Suicide Attempts | 4 weeks
  Whether or not a suicide attempt occurs during the 12-week intervention period will be captured by manual review of electronic health records and the Self-Injurious Thoughts & Behaviors Interview (SITBI).
Number of Suicide Attempts | 8 weeks
  Whether or not a suicide attempt occurs during the 12-week intervention period will be captured by manual review of electronic health records and the Self-Injurious Thoughts & Behaviors Interview (SITBI).
Number of Suicide Attempts | 12 weeks
  Whether or not a suicide attempt occurs during the 12-week intervention period will be captured by manual review of electronic health records and the Self-Injurious Thoughts & Behaviors Interview (SITBI).

SECONDARY OUTCOMES:
Treatment Attendance | 4 weeks, 8 weeks, and 12 weeks
  Treatment attendance during the 12-week intervention period will be captured by manual review of electronic health records and participant-reported outcome survey.
Depressive Symptoms | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Depressive symptoms will be measured using the Patient Health Questionnaire-9 (PHQ-9). The scale values ranges from 0 to 3. Higher total scores mean more severe symptoms.
Intensity of Suicidal Ideation | Baseline, 4 weeks, 8 weeks, and 12 weeks
  The intensity of suicidal ideation will be measured using the Beck Scale for Suicide Ideation (BSS). The scale values ranges from 0 to 2. Higher scores mean more intense suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Smoller, MD, ScD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doupnik SK, Rudd B, Schmutte T, Worsley D, Bowden CF, McCarthy E, Eggan E, Bridge JA, Marcus SC. Association of Suicide Prevention Interventions With Subsequent Suicide Attempts, Linkage to Follow-up Care, and Depression Symptoms for Acute Care Settings: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2020 Oct 1;77(10):1021-1030. doi: 10.1001/jamapsychiatry.2020.1586. PMID 32584936
- [Background] Milner AJ, Carter G, Pirkis J, Robinson J, Spittal MJ. Letters, green cards, telephone calls and postcards: systematic and meta-analytic review of brief contact interventions for reducing self-harm, suicide attempts and suicide. Br J Psychiatry. 2015 Mar;206(3):184-90. doi: 10.1192/bjp.bp.114.147819. PMID 25733570
- [Background] National Action Alliance for Suicide Prevention: Transforming Health Systems Initiative Work Group. Recommended standard care for people with suicide risk: Making health care suicide safe. Education Development Center, Inc. Published online 2018.
- [Background] Office of the Surgeon General (OSG). The Surgeon General's Call to Action to Implement the National Strategy for Suicide Prevention [Internet]. Washington (DC): US Department of Health and Human Services; 2021-. Available from http://www.ncbi.nlm.nih.gov/books/NBK592704/ PMID 37347878